CLINICAL TRIAL: NCT02796287
Title: Longitudinal Monitoring of Cerebral Connectivity 3T MRI in Patients With a Transcient Global Amnesia
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: The principal investigator decided to stop the study.
Sponsor: Fondation Hôpital Saint-Joseph (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: ICTUS
Record Dates: First submitted 2016-06-02; First posted 2016-06-10 (Estimated); Last update posted 2019-02-15 (Actual); Status verified 2018-08

CONDITIONS: Amnesia
Keywords: Amnesia; transient global amnesia
MeSH Terms: conditions — Amnesia; Amnesia, Transient Global

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Patients with Ictus amnesic (Experimental): Patients admitted in the hospital as part of their medical care with amnesic Ictus episode
  Interventions: Procedure: achieving a neuropsychological examination in the acute amnesic phase; Procedure: Neurological consultation with neuropsychological evaluation; Radiation: MRI

INTERVENTIONS:
Procedure: achieving a neuropsychological examination in the acute amnesic phase — achieving a neuropsychological examination in the acute phase in addition to the normal protocole
Procedure: Neurological consultation with neuropsychological evaluation — Neurological consultation with neuropsychological evaluation one year after the acute amnesic phase
Radiation: MRI — Brain MRI with the same protocol or an acquisition time of 15 minutes without gadolinium, one year after the acute amesic phase

SUMMARY:
The transient global amnesia (IA) is defined clinically as a temporary suspension and isolated from the ante and retrograde memory, totally regressing within 24 hours. The causes of AI remain unknown. The diagnosis of IA is based on consensus clinical criteria including the absence of associated location marks. In clinical practice, the MRI is often performed in conjunction with clinical examination because it ensures the absence of differential diagnoses, including stroke.

The visualization of MRI signal abnormalities related to AI directly dependent on the completion time of the review in relation to the onset of symptoms. Typically, no signal abnormality is visible in the hyperacute phase (ie D0-D1) while punctate appear hyperintense on diffusion sequences in hippocampal structures from J2 to J7 to disappear completely. It has been previously demonstrated that the use of higher values of b and / or a better spatial resolution significantly increases the sensitivity of the broadcasting sequence for the detection of these abnormalities hippocampal signal. At St. Joseph Hospital, Investigators explore the AI suspected patients with diffusion tensor sequence (DTI) on our high resolution 3T MRI.

Compared to the classical diffusion sequence, DTI is characterized by the use of a greater number of directions in which the diffusion gradients are applied. One advantage of this technique is to be able to perform tractography of white matter fibers. Thus the "connectome" is a new technique for post-processing of DTI images based tractography and to assess all the networks of nerve fibers in the brain. By this technique, the values of average diffusivity (MD) and fractional anisotropy (FA) can be measured along each of the studied nerve fibers. Group studies thus become feasible to compare quantitatively healthy subjects and patients groups in terms of structural differences within the connectome. The contribution of this technique was recently highlighted in patients with temporal lobe epilepsy.

DETAILED DESCRIPTION:
1. / OBJECTIVES

   The main objective of our study is, using the DTI realized 3T to:

   1.1 Main Objective

   - Highlight changes in brain connectivity induced by the occurrence of transient global amnesia in acute and monitor these remote anomalies (up to 1 year after the initial episode IA).

   1.2 Secondary Objectives
   * Correlate brain connectivity abnormalities identified data of neuropsychological examination
   * Correlate brain connectivity abnormalities identified o Brain morphological data (volumes of gray matter, white matter, hippocampal structures and LCS) o potential hippocampal hyperintensities visible in the acute phase of the diffusion images (number and laterality)

   1.3 Methodology

   DESIGN: biomedical, prospective single-center on topics of AI episode as part of their medical care within the hospital group Paris Saint-Joseph, 185 Rue Raymond Losserand 75014 Paris.

   Study duration: 2 years from May 2015 in the rate of inclusion estimated to average 2-3 patients per month (ie inclusion period of one year: from May 2015 to May 2016 and last follow-up in May 2017 ).

   start and end dates: May 2015 to May 2017 Number of topics to include: This is an exploratory study, single center, on a rare disease, the incidence of stroke is estimated amnesia of 3 to 8 patients per 100 000 per year according to recent studies.
   * Based on a feasibility study previously carried out within the department, Investigators estimate that approximately 30% from refusal to participate in the study.
   * Only 3T MRI allows for the proper sequences: it is only available every other day to practice brain MRI In this context, Investigators therefore believe about 45 the number of subjects may be recruited during the period of inclusion (2 years)
2. / COURSE OF STUDY

   2.1 Patients and MRI

   Only patients referred for achieving their brain MRI as part of a typical transient global amnesia in the Radiology Department of the Paris Saint Joseph Hospital Group will be included in succession.

   For each subject, the following clinical data will be collected:

   - Age, sex
   * Medical background
   * Duration of AI, date and circumstances of occurrence
   * Current Treatments

   In the acute phase, there is no change in the usual care of the patient. The patient has a consultation with a neurologist at D0 / D1 which ensures the typical character of the clinical presentation.

   An MRI is performed on day 2 of the onset of symptoms to confirm the diagnosis.

   The usual course of MRI is not modified in any way, it includes the reception of the patient, information on the MRI scan and search against-indications. The images are acquired using a 3T MRI (GE Discovery MR 750) with 32 elements antenna head. The conventional imaging protocol includes the DTI sequences, FLAIR and 3DT1 without gadolinium (or 15 minutes of acquisition). As part of the study, it is not directed modification of the imaging protocol.

   Changes in the management of patients related to the application of this protocol are:

   - To carry out a neuropsychological examination in the acute phase

   - Renew for one year the episode AI

   o neurological consultation with neuropsychological evaluation

   o brain MRI with the same protocol or an acquisition time of 15 minutes without gadolinium.

   Study design in Annex 2.

   2.1 Post processing

   The post processing of the data will be conducted at the research platform of the Lille University Hospital, which specializes in advanced imaging techniques (Prof. Xavier Leclerc, Mr Renaud Lopes), and include the following steps:
   * From 3D T1 sequence: the parcellation of the cortex regions of interest is necessary for the evaluation of connectome, volume measurements of SG, SB, LCS and seahorses using the software " Freesurfer "
   * From the DTI sequence: obtaining connectivity maps for each subject with measurement of MD and FA
   * Statistical comparison of different groups of subjects (patients vs controls J2 (healthy subjects) patients at 1 year vs controls, patients at Day 2 vs 1 year) and obtaining connectivity graphs showing the significant differences between these groups in terms of FA and MD. The controls (healthy subjects) are obtained from the database "1000 connectomes" available online.
3. / IMAGE ANALYSIS

Image analysis is done in two stages.

1. / interpretation "clinical" images, immediately with the aim to answer the following questions:

   * There is a stroke? another injury? whether the patient is excluded from the study
   * Vascular leukopathy according to the scale of Fazekas? stigmata of ischemic or hemorrhagic lesions?
   * Typical hippocampal hyperintensities AI? laterality and the number of injuries will be collected for each subject.
2. / post processing of images (see above).

4 / STATISTICAL ANALYSIS

* Descriptive analysis of results
* Comparison of connectivity graphs representing the values of FA and MD among the three groups of subjects: normal subjects, patients explored D2, explored patients at 1 year
* SG volume comparison, SB, LCS and seahorses among the three groups of subjects: normal subjects, patients explored D2, explored patients at 1 year
* Search correlation between connectivity and anomalies o 1 / lateral abnormal hippocampal signal,

  * 2 / volumes measured from the sequence and 3DT1
  * 3 / abnormal neuropsychological examination

    5 / ETHICS / REGULATORY:

This protocol presents no added risk to the patient. The initial MRI examination D2 is routinely performed as part of routine monitoring of patients with IA.

Changes in the management of patients related to the application of this protocol is to renew 1-year episode of AI:

* Neurological consultation with neuropsychological evaluation
* Brain MRI with the same protocol as for acute MRI performed an acquisition time of 15 minutes without gadolinium.

Data processing will be carried out within the research platform of the Lille University Hospital of anonymized way. Collaboration is already underway with this research center with several joint publications in the field of inflammatory and vascular diseases. The principal investigator (Dr. Hodel) exercises in both structures.

To start searching the CRC GHPSJ, as a promoter must submit a permit application to the competent authority (ANSM for biomedical research out health product).

In accordance with Article L.1123-6 of the Public Health Code, the research protocol must be submitted by the proponent to the Patient Protection Committee of choice (CPP Ile de France II). The opinion of the committee is notified to the competent authority by the developer before the start of the research.

When the protocol has a quality control of the data by a CRA representative promoter and enters the scope of the CNIL simplified procedure, the developer will ask the head of the computer file (investigator-coordinator research) to commit to compliance with the methodology of reference MR001 simplified.

The inclusion of patients will occur after the patient's information and collection of written consent; its information and consent will be traced in his file.

The patient's consent is sought:

1. / for the use of data acquired in the acute phase for research purposes
2. / to make a new MRI and a consultation of Neurology at 1 year of onset of symptoms

ELIGIBILITY:
Inclusion Criteria:

* Patients with a typical transient global amnesia
* Sent for MRI as part of usual care protocol

Exclusion Criteria:

* Any contraindication of MRI
* Atypical clinical and / or radiological
* Other active disease of the Central Nervous System
* Patients with a history of cerebral infarction

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1 (Actual)
Dates: Start 2015-09-02 (Actual); Primary Completion 2018-12-31 (Actual); Study Completion 2018-12-31 (Actual)

PRIMARY OUTCOMES:
Assessment of change of connectivity graphs representative of the FA (fraction anisotropy) facts | Day 2, 1 year
  Comparison of connectivity graphs representing the FA values between the three groups of subjects : normal subjects , patients explored J2, explored patients at 1 year
Assessment of change of connectivity graphs representative of the MD (mean diffusivity) facts | Day 2, 1 year
  Comparison of connectivity graphs representing the MD values between the three groups of subjects : normal subjects , patients explored J2, explored patients at 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Jerome HODEL, MD, Principal Investigator — Fondation Hôpital Saint-Joseph
Locations (1):
- Groupe Hopitalier Paris Saint Joseph Service de radiologie, Paris, Île-de-France Region, France